CLINICAL TRIAL: NCT02052921
Title: Open Randomized Study of Observation Versus Surgical Resection in Patients With Rectal Cancer Who Achieved Complete Clinical Response After Neoadjuvant Chemoradiotherapy
Brief Title: Observation Versus Surgical Resection in Patients With Rectal Cancer Who Achieved Complete Clinical Response After Neoadjuvant Chemoradiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: During the execution time foreseen in the project, the expected number of patients was not reached.
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP172/11
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: Observation; Rectal Resection; complete clinical response; neoadjuvant chemoradiotherapy.
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectal resection (Active Comparator): Surgical rectal resection
  Interventions: Procedure: Rectal resection
- Observation (Experimental): Conservative approach
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: Rectal resection — Surgical rectal resection
  Arms: Rectal resection
Other: Observation
  Arms: Observation

SUMMARY:
With the possibility of pathological complete response in surgical specimens, some authors have proposed non-operative management of the patient group, when re-staged after neoadjuvant treatment, have complete clinical response. So far, this approach remains discussed in the literature, and there are still many uncertainties that patients with clinical complete response after chemoradiotherapy in fact no detectable viable tumor and may be omitted of radical surgical treatment. It is a still investigational approach and actually gained space even for patients with very high or who refuse surgery after all clarifications surgical risk.

Hypothesis: The preservation of the rectum in patients with adenocarcinoma of the middle and distal rectum (up to 10 cm) reaching clinical complete response after neoadjuvant chemoradiotherapy have similar rate of the rectal cancer recurrence than patients who underwent surgical rectal resection.

This will be a prospective, randomized, open label phase II of surgical resection versus conservative treatment (observation) in patients with mid and distal rectal cancer who achieved complete after neoadjuvant chemoradiotherapy combined with clinical response.

The main objective of this study is to assess whether conservative approach is similar to rectosigmoidectomy with complete mesorectal excision or amputation abdminoperineal the rectum in patients with complete clinical response after neoadjuvant therapy combined chemoradiotherapy.

Patient Selection: To be eligible patients who have neoadjuvant prior histologic diagnosis of rectal adenocarcinoma, tumors located within 10 cm from the anal verge, a complete clinical response after treatment with chemoradiotherapy for rectal tumors staged clinical and radiological T3-4 N0 M0 or T (any) N + M0, absence of colorectal synchronous tumors.

Treatment: Eligible patients will be randomized 1:1 to resection of the rectum or notice. The period for randomization of patients will be 12 weeks after the last dose of radiotherapy / chemotherapy, so that we can properly assess the antitumor response as described above. After randomization, patients in the surgical group will undergo resection of the rectum with complete excision of mesorectal within 2 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of rectal adenocarcinoma
* tumors located within 10 cm from the anal verge by rigid proctoscopy measurement
* Complete clinical response after neoadjuvant treatment with chemoradiotherapy for rectal tumors clinical and radiologically staged as T3-4 N0 M0 or T (any) N + M0
* Absence of colorectal synchronous tumors
* Age between 18 and 75 years
* ECOG performance scale ≤ 2,
* last dose of chemotherapy / radiation therapy in up to 12 weeks
* Good organic function
* Absence of serious comorbidities defined by the doctor to prevent surgical resection of the rectum and / or neoadjuvant therapy.

Exclusion Criteria:

* Comorbidities clinically significant where surgical resection and / or neoadjuvant therapy is impossible, according to medical assessment.
* Prior antineoplastic therapy different from neoadjuvant therapy.
* History of Crohn's disease or ulcerative colitis.
* Confirmation or strongly suspected inherited polyp syndrome.
* Pregnant women or during lactation (women of childbearing age should have a negative pregnancy test).
* Concurrent participation in another research protocol involving therapeutic intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years

SECONDARY OUTCOMES:
Operative complication rate | 30 days

OTHER OUTCOMES:
Presence of viable tumor in the surgical specimen | 3 years
Pattern of recurrence | 3 years
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cecconello, MD, Principal Investigator — Faculdade de Medicina da USP; Ulysses Ribeiro, MD, Study Director — Instituto do Câncer do Estado de São Paulo
Locations (1):
- Instituto Do Câncer Do Estado de São Paulo, São Paulo, Brazil